CLINICAL TRIAL: NCT05534828
Title: Risk Factors for the Occurrence of Post Intensive Care Syndrome (PICS) At 3 Months After a Stay in the Rangueil Multipurpose Resuscitation Unit of the Toulouse University Hospital
Brief Title: Risk Factors for the Occurrence of Post Intensive Care Syndrome (PICS)
Acronym: PICS3
Status: Completed | Type: Observational
Sponsor: University Hospital, Toulouse (Other)
Responsible Party: Sponsor
Other Study IDs: RC31/22/0215; 2022-A01371-42 (Other: ID-RCB)
Record Dates: First submitted 2022-09-06; First posted 2022-09-10 (Actual); Last update posted 2024-09-25 (Actual); Status verified 2024-09

CONDITIONS: Post Intensive Care Syndrome
MeSH Terms: conditions — postintensive care syndrome

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

INTERVENTIONS:
Diagnostic Test: A consultation — A consultation at three months of discharge from the intensive care unit in the population of patients surviving a multivalent intensive care unit stay

SUMMARY:
Monocentric, observational, descriptive RIPH3 study with prospective data collection.

DETAILED DESCRIPTION:
A consultation in the form of a teleconsultation with video conference is proposed to all adult patients who have stayed more than 24 hours in the Rangueil intensive care unit.

This consultation is scheduled and will take place approximately three months after the end of the stay in the intensive care unit.

During this consultation, signs will be sought through questioning to detect or even diagnose the presence of a PICS.

We will also look for elements that will allow us to characterize people with CHIP.

If a PICS was detected during the consultation, the summary letter sent to the attending physician informs him/her of

1. The presence of a CHIP in his patient
2. The nature of this CHIP (CHIP with a purely psychological component, CHIP with a psychological and physical component, etc.) In this same summary letter, the attending physician will be offered a list of specialists practicing at the CHU who are likely to take charge of the patient's CHIP.

ELIGIBILITY:
Inclusion Criteria:

* adult patient
* hospitalized in the intensive care unit of Rangueil of the TOULOUSE University Hospital
* length of stay in intensive care equal or superior to 24 hours
* affiliated to a social security system
* having expressed no objection to participate in the study

Exclusion Criteria:

* minor patient
* no consent to the study
* patient not capable of expressing his "non opposition" to the study
* patient under guardianship, curatorship or safeguard of justice

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: population of patients surviving a stay in polyvalent resuscitation
Sampling Method: Probability Sample
Enrollment: 97 (Actual)
Dates: Start 2022-10-10 (Actual); Primary Completion 2023-06-30 (Actual); Study Completion 2023-06-30 (Actual)

PRIMARY OUTCOMES:
Incidence at 3 months of PICS | month 3
  Incidence at 3 months of PICS as defined below:
  A PICS is defined as ''present'' at the 3-month visit if the patient has one or more of the following:
  * Impaired quality of life as defined by a 5D5L EQ score greater than or equal to 3 on at least 1 dimension of the questionnaire.
  * Anxiety symptoms defined by a HADS anxiety score greater than or equal to 11.
  * Depressive symptoms defined by a HADS depression score greater than or equal to 11.
  * Symptoms of post-traumatic stress defined by a PCL 5 score greater than or equal to 33.
  * Symptoms of undernutrition defined by an NRS score greater than or equal to 3.
  * Pain symptoms defined by a DN4 score greater than or equal to 4 and/or an EVS score greater than or equal to 4.

CONTACTS AND LOCATIONS:
Locations (1):
- University Hospital of Toulouse, Toulouse, France

IPD SHARING:
Plan to Share IPD: No